CLINICAL TRIAL: NCT02733887
Title: Research on the Lymphoma Staging and Therapeutic Evaluation of 18F-FDG PET/CT Comparing With Whole Body MRI IVIM Functional Imaging
Brief Title: MRI Compared to PET/CT for Staging and Treatment Response in Lymphoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangxi Medical University (Other)
Responsible Party: Principal Investigator, Chengcheng Liao, Director, Principal Investigator, Clinical Professor, Guangxi Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PET-MRI/lymphoma
Record Dates: First submitted 2016-03-17; First posted 2016-04-12 (Estimated); Last update posted 2016-04-12 (Estimated); Status verified 2016-04

CONDITIONS: Lymphoma
MeSH Terms: conditions — Lymphoma | interventions — Magnetic Resonance Imaging; Positron Emission Tomography Computed Tomography; Fluorodeoxyglucose F18

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- lymphoma (Experimental): The lymph nodes or masses, fludeoxyglucose F18 positron emission tomography/computed tomography(PET/CT) standard uptake value(SUV) results, whole body magnetic resonance imaging(MRI) intravoxel incoherent motion(IVIM) sequence D, D*,f values and MRI volumes of lymphoma were compared before and after the chemotherapy in this project prospectively to provide data for evaluating the dependency and differences of PET/CT and whole body MRI in lymphoma staging and therapeutic evaluation.
  Interventions: Device: magnetic resonance imaging; Device: positron emission tomography/computed tomography; Radiation: fludeoxyglucose F 18

INTERVENTIONS:
Device: magnetic resonance imaging — MRI was performed on a 3 Tesla system (GE Discovery 750W). A single-shot,echo-planar imaging-based, spectral adiabatic inversion recovery DWI sequence was obtained with b values of 0,30,50,80,100,150,200,400,600,800 and 1,000.
  Other Names: MRI
Device: positron emission tomography/computed tomography — 18F-FDG-PET/CT was performed using a multidetector PET/CT system (GE Discovery ST16). Patients fasted for 6 hours before imaging.
  Other Names: PET/CT
Radiation: fludeoxyglucose F 18 — Patients fasted for 6 h before receiving FDG intravenously. A dose of 5.18-7.4 MBq/kg was used.
  Other Names: 18F-FDG; FDG

SUMMARY:
The lymph nodes or masses,positron emission tomography/computed tomography (PET/CT) standardized uptake values(SUV) results, whole body magnetic resonance imaging(MRI) intravoxel incoherent motion(IVIM) sequence D, D*, f values and MRI volumes of lymphoma patients were compared before and after the chemotherapy in this project prospectively to provide data for evaluating the dependency and differences of PET/CT and whole body MRI in lymphoma staging and therapeutic evaluation. Long-term therapeutic effect indexes obtained in follow-up visits of patients such as Overall Survival(OS), Progression Free Survival (PFS) etc. were used to evaluate the diagnostic sensitivity and differences of MRI and PET/CT. The research could provide a new method of nonionizing radiation iconography for physicians to give appropriate treatments and predict prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Lymphoma subtypes were diagnosed on the basis of tissue samples obtained by biopsy or surgery according to the criteria outlined in the current World Health Organization (WHO) classification of hematologic and lymphoid malignancies, by a reference pathologist.
* Patients who gave written informed consent were referred for DWI-MRI and 18F-FDG-PET/CT.
* Stable physical medical conditions (patients conscious and comfortable, scheduled for an elective diagnostic imaging).

Exclusion Criteria:

* Pregnancy, general contraindications to MRI, and therapeutic interventions between DWI-MRI and 18F-FDG-PET/CT were used.

Ages: 8 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2016-02; Primary Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
18F-FDG uptake in lymphomas with PET/CT | Within 30 days prior to start of chemotherapy
  Different 18F-FDG uptake values in lymphoma tissue (e.g. SUVmax, SUVmean, binding potential) will be measured and correlated with immunohistochemically determined somatostatin receptor status, lymphoma aggressiveness and tissue biomarkers
Agreement between DWI-MRI and 18F-FDG PET/CT at diagnosis | Within 30 days prior to start of chemotherapy
  Region based agreement (%; kappa value) of DWI-MRI with 18F-FDG PET/CT at diagnosis.
Agreement between DWI-MRI and 18F-FDG PET/CT in follow-up examinations | 2 weeks after the 4th cycle of chemotherapy
  Region based agreement (%; kappa value) of DWI-MRI with 18F-FDG PET/CT after completion of chemotherapy for treatment response assessment

SECONDARY OUTCOMES:
Overall Survival | 12 months
Progression Free Survival | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Tumor Hospital，Guangxi Medical University, Nanning, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cheson BD, Fisher RI, Barrington SF, Cavalli F, Schwartz LH, Zucca E, Lister TA; Alliance, Australasian Leukaemia and Lymphoma Group; Eastern Cooperative Oncology Group; European Mantle Cell Lymphoma Consortium; Italian Lymphoma Foundation; European Organisation for Research; Treatment of Cancer/Dutch Hemato-Oncology Group; Grupo Espanol de Medula Osea; German High-Grade Lymphoma Study Group; German Hodgkin's Study Group; Japanese Lymphorra Study Group; Lymphoma Study Association; NCIC Clinical Trials Group; Nordic Lymphoma Study Group; Southwest Oncology Group; United Kingdom National Cancer Research Institute. Recommendations for initial evaluation, staging, and response assessment of Hodgkin and non-Hodgkin lymphoma: the Lugano classification. J Clin Oncol. 2014 Sep 20;32(27):3059-68. doi: 10.1200/JCO.2013.54.8800. PMID 25113753